CLINICAL TRIAL: NCT07299851
Title: Randomized, Double-blind, Placebo-controlled Study With 12 Weeks Oral Supplementation With a Formulation Based on Cetylated Fatty Acids to Support the Early Stage of Long Lower Limb Bone Healing After Fracture Stabilization
Brief Title: Oral Supplementation With a Formulation Based on Cetylated Fatty Acids for Post-fracture Long Bone Healing
Acronym: CETIULTRA-BONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanutra S.p.a. (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CETI ULTRA-BONE
Record Dates: First submitted 2025-11-17; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Fracture Femur; Fracture Tibia
MeSH Terms: conditions — Femoral Fractures; Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFA-based supplement group (Experimental): Participants will orally consume the assigned product for at least 12 weeks. Intake will be initiated from the day of Baseline (Visit 0) after all study procedures being performed until the morning of the last visit (Visit 3).
  Participants will take 2 sachets a day directly in their mouth.
  Interventions: Dietary Supplement: CFA-based food supplement
- Placebo group (Placebo Comparator): Participants will orally consume the assigned product for at least 12 weeks. Intake will be initiated from the day of Baseline (Visit 0) after all study procedures being performed until the morning of the last visit (Visit 3).
  Participants will take 2 sachets a day directly in their mouth.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CFA-based food supplement — oral gel containing cetilated fatty acids
  Arms: CFA-based supplement group
Other: Placebo — oral gel coloured and flavoured as the IP
  Arms: Placebo group

SUMMARY:
This clinical study aims to evaluate the potential benefits of a formulation based on Cetylated Fatty Acids in improving fracture healing of long bones in the lower limbs. The investigational product is administered orally over a 12-week period. Study procedures are limited to standard imaging techniques (radiography and echography), blood sampling, and completion of validated quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 85 years old
* Presence of simple closed unifocal fracture (transverse, oblique, spiral, butterfly-shaped) in a long bone which need a standard of care surgical stabilization
* Presence of diaphyseal fracture of lower limb (femur or tibia, Subtrochanteric fracture are also allowed)
* Presence intramedullary nail
* Weight bearing as tolerated after surgery
* Having signed an informed consent, understand study procedures and ability to follow them
* Agreed to stop vitamin D intake for participants who take prophylactic Vitamin D

Exclusion Criteria:

* Treatment with vitamin D for medical purpose (Non-union, osteoporosis…)
* BMI > 30
* Open fracture
* Intra articular fracture
* Metaphyseal fracture
* Polytrauma patient (injury severity score: ISS >= 16)
* More than one lower limb long bone fracture
* Bridging plate
* Fracture treated conservatively with plaster
* Presence of active infection (body temperature ≥ 38°C or other symptoms)
* Any sign of severe vascular compromise across the fracture site (such as compartment syndrome, presence of serious vascular damage, etc.)
* Pathological fracture or diseases with a risk of recurrent falling (e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope)
* Participants with known bone disease which would negatively impact on the bone healing process
* Participants currently being treated with radiation, chemotherapy, immunosuppression, or steroid therapy
* Diabetic participants
* Daily smoker participants (cigarette or vaping containing nicotine)
* Participants under cortisone intake
* Participants under rheumatic medications intake
* Allergy or adverse effect of food supplement composition
* Unwilling or unable to take study medication
* Chronic drug or alcohol abuse
* Pregnant or breastfeeding at the time of enrolment
* Any other investigational treatment or food supplement within 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment of Callus Formation using the modified Radiographic Union Score for Tibia (mRUST). | 6 weeks after fracture stabilization
  Comparison between groups of radiographic assessment of the callus formation using mRUST 6 weeks after fracture stabilisation. The mRUST scale ranges from 4 to 16 points, where higher scores indicate better fracture healing (greater callus formation and union).

SECONDARY OUTCOMES:
Pain Assessment at Fracture Site using the Visual Analog Scale (VAS) | 4 weeks after fracture stabilization
  Change from baseline in pain perception in clinical assessment using the VAS 4 weeks after fracture stabilization. The VAS ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse outcomes (greater pain intensity).
Ultrasonographic Assessment of Callus Formation | 4 weeks after fracture stabilization
  Change from placebo group in ultrasonographic evaluation of hypervascularisation and callus formation. Measurement of callus size (length and thickness) in millimeters using B-mode ultrasound imaging at the fracture site. The assessment is performed 4 weeks after fracture stabilization. Larger callus size indicates better bone healing.
Radiographic Assessment of Callus Formation (modified Radiographic Union Score for Tibia - mRUST) | 12 weeks after fracture stabilization
  Radiographic union will be evaluated using the modified Radiographic Union Score for Tibia (mRUST), which rates healing on a 4-16 scale, with higher scores indicating better callus formation and more advanced fracture healing. Comparison between groups at Week 12.
Pain Assessment at Fracture Site (Visual Analog Scale - VAS) | 12 weeks after fracture stabilization
  Pain at the fracture site will be assessed using the Visual Analog Scale (VAS), a 0-100 mm scale, where higher scores indicate worse pain. The endpoint evaluates the change from baseline to Week 12.
Incidence of Complications | 4 weeks and 12 weeks after fracture stabilization
  Comparison between groups of the number of complications observed at 4 and 12 weeks after fracture stabilization. Complications include superficial infection, deep infection, wound breakage, failure of fixation, bleeding, severe blood loss, nerve damage, swelling, deep vein thrombosis, and delayed healing.
Minimal Clinically Important Improvement (MCII) | 4 weeks and 12 weeks after fracture stabilization
  The MCII is calculated using the Visual Analog Scale (VAS) for pain, a 0-100 mm scale where higher scores indicate worse pain. MCII is defined as an absolute improvement of ≥15 mm or a relative improvement of ≥20% from baseline. The measure represents the proportion of participants achieving clinically meaningful pain improvement at each time point.
Participant Acceptable Symptom State (PASS) | 4 weeks and 12 weeks after fracture stabilization
  PASS is determined using the Visual Analog Scale (VAS) for pain, a 0-100 mm scale where higher scores indicate worse pain. PASS is defined as achieving a pain score <30 mm, corresponding to a symptom state considered acceptable by the participant. The measure represents the proportion of participants reaching this threshold.
Participant Global Assessment (PGA) | 4 weeks and 12 weeks after fracture stabilization
  PGA is assessed using a Visual Analog Scale (VAS), a 0-100 mm scale where higher scores indicate worse overall perception of recovery. Participants rate their overall status, taking into account pain, function, and wellbeing. Between-group comparison will be performed at each time point.
Lower Extremity Functional Scale (LEFS) | 4 weeks and 12 weeks after fracture stabilization
  Lower-limb functional recovery will be assessed using the Lower Extremity Functional Scale (LEFS), a validated 20-item questionnaire where each item is scored on a 0-4 scale. Total scores range from 0 to 80, with higher scores indicating better lower-extremity function. Between-group comparison will be performed at each visit.
Quality of Life using the Short Form-36 (SF-36) questionnaire. | 4 weeks and 12 weeks after fracture stabilization
  Health-related quality of life will be assessed using the Short Form-36 (SF-36) questionnaire. The SF-36 includes 8 domains, each scored from 0 to 100, where higher scores indicate better health status. Summary and domain-level results will be compared between groups at each time point.
Painkiller and NSAID Consumption | 4 weeks and 12 weeks after fracture stabilization
  Comparison between groups of the number of painkillers and NSAIDs consumed.
Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) | 4 weeks and 12 weeks after fracture stabilization
  Comparison of the number of adverse events and serious adverse events reported.
Participant Compliance Rate | 4 weeks and 12 weeks after fracture stabilization
  Comparison between groups of participant compliance with study product intake
Participant Satisfaction | 4 weeks and 12 weeks after fracture stabilization
  Participant satisfaction with the study product will be assessed using a Likert scale, ranging from 1 to 5, where higher scores indicate greater satisfaction. The measure evaluates the participant's subjective perception of the product's acceptability and overall experience with the supplementation regimen. Comparison between groups will be performed at each study visit where data are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Meirhaeghe, Principal Investigator — Department of Orthopaedics and Traumatology Ghent University Hospital (UZ Gent), Belgium
Locations (6):
- Belgium (6):
  - AZ Monica, Deurne, Antwerp
  - Algemeen Ziekenhuis Herentals, Herentals, Antwerp
  - Hôpital Erasme - Cliniques Universitaires de Bruxelles, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel, Brussels, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent, Flanders
  - Ziekenhuis Oost-Limburg, Genk, Limburg

IPD SHARING:
Plan to Share IPD: No